CLINICAL TRIAL: NCT05460741
Title: Effects of Integrated Exercise Approach on Strength, Postural Stability and Biomarkers of Menstrual Cycle in Eumenorrheic Females
Brief Title: Integrated Exercise Approach Strength Postural Stability Menstrual Cycle Biomarkers Eumenorrheic Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Collaborators: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC/Lhr/22/1101
Record Dates: First submitted 2022-05-31; First posted 2022-07-15 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Females; Menstrual Discomfort
Keywords: exercise performance; menstrual cycle; sex steroid hormones

STUDY DESIGN:
Intervention Model Description: there will be 2 groups. one will be given the education related to menstrual cycle and other will be given intervention along with education. then the outcomes will be assessed at multiple times of study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- integrated exercise approach (Experimental): an integrated exercise will be used which is the exercise plan that will be formulated using strengthening and endurance exercises.
  Interventions: Other: integrated exercise approach
- eumenhorreic females (Experimental): strength, postural stability and biomarkers of menstrual cycle in eumenhorreic females.
  Interventions: Other: educational program

INTERVENTIONS:
Other: integrated exercise approach — Integrated exercise plan will be given for 16 weeks with frequency of 3 times per week, with duration of session to be 50 minutes being 30 minutes of exercise in total and 10 minutes of rest and 10 min of warm up and cool down exercises.
  Other Names: educational program
  Arms: integrated exercise approach
Other: educational program — educational program related to menstrual cycle will be given to females.
  Arms: eumenhorreic females

SUMMARY:
The study will determine the effects of integrated exercise approach on strength, postural stability and biomarkers (estrogen, progesterone and testosterone) of menstrual cycle in eumenorrheic females and translation of Unified Balance Scale will be done.

DETAILED DESCRIPTION:
In 2021, a study was conducted in which evaluation of the effects of phases of menstrual cycles on the performance of athletes was done. It was concluded that the performance of athletes is effected along with phases of MC with strength and aerobic performance being effected during late luteal phase and anerobic performance was reduced during late follicular phase.

In 2021, another study was conducted. The bidirectional interactions between the menstrual cycle, exercise training and macronutrient intake in women was studied. It was concluded in their study that exercise interventions have an effect on the hormonal level and in turn their physical activity but it varies so much from one women to other that no generalization may be made and need to be investigated more.

In 2020, a systematic review related to effects of menstrual cycle phase on exercise performance in eumenorrhic women was done. It was concluded that exercise performance may get reduced in the early follicular phase so the practitioners working with sportswomen must consider the phases of their menstrual cycle and look for the potential times when their performances may be enhanced that is in all phases except follicular phase to get the optimum results during their games.

In 2020, the study related to the effects of sex steroids on joint position sense during different phases of menstrual cycle was done. It was concluded in this study that in early follicular phase as the levels of sex steroid hormone specifically oestrogen is low, it leads to decrease joint position sense as compared to luteal and ovulatory phases where there is less error in joint position sense. These findings are more pronounced in the hip joint due to greater motor neuron activity of these muscles.

In 2019, study was conducted in which it was documented that when exercise is performed it has certain physiological effects and the phases of menstrual cycle plays an important role in modulating these physiological responses during recovery phase. He postulated that a more robust recovery CK and IL-6 response occur in the MF of the menstrual late cycle when female sex hormones are reduced.

In 2018, the combined effects of strength and endurance training on the biomarkers and physical activity of healthy women were studied. It was hypothesized by this study that even with limited exposure to strengthening and endurance programs the females can get benefit as compared to the sedentary women. Their health biomarkers also showed positive effects.

In 2017, evaluation of muscle strength variations and also the rate of fatigue during various phases of the menstrual cycle in young adults was done. It was hypothesized that cyclical variation in endogenous reproductive hormones increases the muscle strength in follicular phase of the menstrual cycle. Thus provide support for the influence of these hormones in regulation of these parameters in the premenopausal age group.

In 2017, study was conducted to see the effects of menstrual cycle phases on the performance of athletes specifically soccer players. The result of this study was in support of reduction in maximal endurance performance during the mid luteal phase of the menstrual cycle confirming the fact that the phases of menstrual cycle do have effect on the endurance of the athletes so the trainer should consider these fact while training of the female athletes.

In 2015, a systematic review was done to include 40 studies in which different exercises were done including strength exercises, endurance exercises and free style exercises and their effects were then seen on sex hormones. It was concluded by this study that physical activity which ever type it may be induces a decrease in circulating sex hormones and this induces the beneficial effects on women. It also helps in weight loss and overall physical well being.

So it is evident that some work has been done on documenting the effects of exercise on estrogen, progesterone level but little is known about the effects of exercise on testosterone levels. The regulation of both of them is necessary to maintain the effective force production of muscles, joint laxity and balance control. Moreover, there is no single generalized approach which focuses on strength, postural stability and postulated to effects hormones.

ELIGIBILITY:
Inclusion Criteria:

* Females between the ages of 18 to 40 years.
* Females having BMI between 18.5 to 24.9 (normal)
* Females being able to maintain sitting balance independently without using upper limbs or having score of 25 on trunk control test.

Exclusion Criteria:

* Females having oral contraceptives.
* Females who are pregnant.
* Females who have any menstruation issues like endometriosis, ovarian cysts etc
* Females who have c section 6 months ago.
* Females who are lactating.
* Females having other co morbidities like cardiac event, seizures, any injury that will affect the study.
* Females having history of fall 6 months ago.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — females having no problem in menstrual cycle
Enrollment: 60 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
ELISA | 4 months
  progesterone, testosterone and estrogen of the females with no menstrual cycle dysfunction will be documented at baseline and then the exercise plan along with menstrual cycle education will be given to one group and just educational program will be given to other. the biomarkers will then be assesd after 2 months and at the end of study i.e, after 4 months.The unit of measurement of progesterone is ng/ml. progesterone is less than 1.5ng/ml in follicular phase, greater than 3ng/ml in ovulatory phase and 2 to 25ng/ml in luteal phase, testosterone is measured in nmol/L, being 0.32nmol/L in follicular phase and 0.35nmol/L in ovulatory and luteal phase. estrogen measured in pg/ml, being less than 50pg/ml in follicular phase, 400 pg/ml in ovulatory phase and upto 200pg/ml in luteal phase.this test has 68% sensitivity and 98% specificity

SECONDARY OUTCOMES:
hand held dynamometer | 4 months
  grip strength of females will be taken at baseline and then after 2 months and 4 months to see the effect of intervention on it. It ranges from 21.5 kg to 35.3kg which varies from dominant to non dominant hand and varies with age too. it has high reliability from 0.85 to 0.99
pressure biofeedback unit | 4 months
  it will be used to measure the strength of lower limb at baseline, after 2months and 4 months. For quadriceps it ranges from 16 to 20 kg and 18 to 20 kg in hamstrings. This test has a reliability of 0.86

OTHER OUTCOMES:
global postural system | 4 months
  it is a software that is used to check the postural stability, evaluating the postural sway which will be checked at baseline, 2 months and 4 months. The normal values for postural sway in sagittal plane is 12mm whearas in frontal plane it is 8.17mm. This test has the reliability of 0.38

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, phd*, Principal Investigator — Riphah International University
Locations (1):
- Society, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rocha-Rodrigues S, Sousa M, Lourenco Reis P, Leao C, Cardoso-Marinho B, Massada M, Afonso J. Bidirectional Interactions between the Menstrual Cycle, Exercise Training, and Macronutrient Intake in Women: A Review. Nutrients. 2021 Jan 29;13(2):438. doi: 10.3390/nu13020438. PMID 33572821
- [Background] Kitajima Y, Ono Y. Estrogens maintain skeletal muscle and satellite cell functions. J Endocrinol. 2016 Jun;229(3):267-75. doi: 10.1530/JOE-15-0476. Epub 2016 Apr 5. PMID 27048232
- [Background] Le J, Thomas N, Gurvich C. Cognition, The Menstrual Cycle, and Premenstrual Disorders: A Review. Brain Sci. 2020 Mar 27;10(4):198. doi: 10.3390/brainsci10040198. PMID 32230889
- [Background] Smith MJ, Adams LF, Schmidt PJ, Rubinow DR, Wassermann EM. Effects of ovarian hormones on human cortical excitability. Ann Neurol. 2002 May;51(5):599-603. doi: 10.1002/ana.10180. PMID 12112106
- [Derived] Shahid W, Noor R. Effects of integrated exercise approach on total testosterone levels in eumenorrheic women: a randomized controlled trial. Sci Rep. 2025 May 5;15(1):15692. doi: 10.1038/s41598-025-00599-x. PMID 40325081
- [Derived] Shahid W, Noor R. Impact of BRACTS exercises on muscular strength in eumenorrheic women. Sci Rep. 2025 Feb 5;15(1):4430. doi: 10.1038/s41598-025-87352-6. PMID 39910068